CLINICAL TRIAL: NCT01848509
Title: A Telemedicine System for the Follow-up of Patients With SAS
Brief Title: Telemedicine for Sleep Apnea Patients
Acronym: Respir@dom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012-A00713-40; K120501 (Other: APHP - Clinical research department)
Record Dates: First submitted 2013-04-10; First posted 2013-05-07 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Sleep Apnea
Keywords: CPAP; adherence; SAOS; telemedicine
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without telemonitoring (No Intervention): Without teletransmission of alerts
- With telemonitoring (Experimental): With teletransmission of alerts
  Interventions: Device: With teletransmission

INTERVENTIONS:
Device: With teletransmission — Teletransmission of alerts
  Arms: With telemonitoring

SUMMARY:
Objective: Set up an interoperable telemedicine system for the follow-up of patients with sleep apnea syndrome.

DETAILED DESCRIPTION:
The medico-economics protocol will use the MAST (Methodology for Assessment of Telemedicine) criteria. 200 patients will be randomized into 2 arms (telemedicine with GPRS transmission of CPAP data from patients' home and classical follow-up) during the 3 first months of the follow-up. The main end-point is CPAP compliance with the aim of detecting a mean increase of at least 1hr in the use of CPAP.

ELIGIBILITY:
Inclusion Criteria:

* AHI > 30/hr
* hypersomnolence
* agreement for the use of CPAP
* internet and GSM connection

Exclusion Criteria:

* central apnea >20%,
* pneumothorax,
* severe nasal obstruction,
* previous pharyngeal surgery,
* severe COPD,
* heart failure,
* previous use of CPAP,
* no social security coverage,
* unavailability,
* no GSM and internet network

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
CPAP adherence measured by the number of hours of nightly use | 3 Months

SECONDARY OUTCOMES:
economics: cost estimation: investment and running costs | 3 months
Quality of life | 3 months
  SF36 (french version) and FOSQ (Functional Outcomes of Sleep Questionnaire)
Organizational changes of home care providers and medical structures | 9 months after the first patient inclusion
Perception of healthcare professionals (autoquestionnaire RENEWING HEALTH) | 3 months
Patients satisfaction | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ESCOURROU, MD, PhD, Principal Investigator — AP-HP - Antoine Béclère Hospital
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Béclère Hospital, Clamart, France